CLINICAL TRIAL: NCT04593251
Title: A Multicentre, SAD, and MAD Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IV Treatment of CALY-002 in Healthy Subjects and Subjects With Celiac Disease and Eosinophilic Esophagitis
Brief Title: Dose Escalation Study to Evaluate an Experimental New Treatment (CALY-002) in Healthy Subjects and Subjects With Celiac Disease and Eosinophilic Esophagitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calypso Biotech BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CALY-CL19-001
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Eosinophilic Esophagitis; Celiac Disease
Keywords: anti IL-15; CalypsoBiotech; Calypso Biotech; Celiac Disease; Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis; Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CALY-002 (Experimental)
  Interventions: Biological: CALY-002
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CALY-002 — 1-hour intravenous infusion
  Arms: CALY-002
Biological: Placebo — 1-hour intravenous infusion
  Arms: Placebo

SUMMARY:
This is a single and multiple ascending study to characterize the safety, PK, PD and clinical effect in healthy volunteers and participants with Celiac Disease and Eosinophilic Esophagitis.

DETAILED DESCRIPTION:
This is a multi-site, randomized, placebo controlled single and multiple dose escalation study of an anti-IL-15 mAb (CALY-002). The study initiates as placebo controlled, randomized trial with a single ascending dosing part in healthy subjects and commences with a multiple ascending dosing part in participants with Celiac Disease undergoing a gluten challenge and includes open label multiple dose expansion cohorts in participants with Eosinophilic Esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Part A. Healthy Subjects:

  1. Male or female aged between 18 and 50 years (both inclusive)
  2. Must be healthy on the basis of the physical examination findings, clinical laboratory tests, medical history, vital signs, and cardiac monitoring (normal 12 lead electrocardiogram [ECG] results) performed at screening, in the opinion of the investigator
* Part B. Subjects with Celiac Disease (CeD):

  1. Male or female ≥ 18 years of age.
  2. Diagnosis of CeD by intestinal biopsy at least 12 months prior to screening as confirmed by medical records.
  3. No histological signs of active CeD at screening
  4. Gluten-free diet (GFD) for at least 12 consecutive months prior to screening
  5. Willing to undertake a gluten challenge (intake of approximately 3 g of gluten daily) for 56 consecutive days
  6. Must be healthy on the basis of physical examination findings, clinical laboratory tests, medical history, vital signs, and cardiac monitoring (normal 12 lead ECG results) performed at screening, in the opinion of the investigator.
* Part C. Subjects with Eosinophilic Esophagitis (EoE):

  1. Male or female ≥ 18 years of age.
  2. Must have endoscopically confirmed and documented diagnosis of EoE
  3. Should exhibit active symptoms of dysphagia with more than 3 episodes of dysphagia during a period of 2 weeks during screening.
  4. Must have clinically active disease
  5. Must have had a relapsed EoE or did not respond after first line therapy
  6. Subject must be healthy on the basis of physical examination findings, clinical laboratory tests, medical history, vital signs, and cardiac monitoring (normal 12 lead ECG results) performed at screening, in the opinion of the investigator.

Exclusion Criteria:

* Part A. Healthy Subjects excluded:

  1. Any significant medical condition, laboratory abnormality, or psychiatric illness
  2. Any condition that confounds the ability to interpret data from the study.
  3. Currently receiving or has been previously treated with a biologic agent.
  4. History of anaphylactic reactions to protein therapeutics.
  5. Has current or recent (within 4 weeks prior to screening) signs or symptoms of infection that require parenteral antibiotic administration.
  6. Has evidence of SARS-CoV-2 infection and/or subject Is deemed at risk for the coronavirus disease (COVID-19)
  7. Has had major surgery (including joint surgery) within 8 weeks prior to screening and hospitalisation for a clinically relevant event within the 4 weeks prior to screening.
* Part B. Subjects with Celiac Disease (CeD) excluded:

  1. A concurrent active autoimmune disease (other than CeD) that requires systematic treatment with immunosuppressants.
  2. Has severe complication of CeD such as refractory CeD.
  3. Has active (microscopic) colitis with clinical signs of diarrhoea and abdominal pain.
  4. Is currently receiving or has been previously treated with a biologic agent.
  5. Has a history of anaphylactic reactions to protein therapeutics.
  6. Subject has evidence of SARS-CoV-2 infection and/or subject is deemed at risk for the coronavirus disease (COVID-19).
* Part C: Subjects with Eosinophilic Esophagitis (EoE) excluded:

  1. Has a hyper-eosinophilic syndrome.
  2. Has a concurrent active autoimmune disease (other than EoE) that requires treatment with immunosuppressants.
  3. Has active (microscopic) colitis with clinical signs of diarrhoea and abdominal pain.
  4. Currently receiving or has been previously treated with a biologic agent.
  5. Has a history of anaphylactic reactions to protein therapeutics.
  6. Subject has evidence of SARS-CoV-2 infection and/or subject is deemed at risk for the coronavirus disease (COVID-19).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse event | through study completion, an average of 3 months post last dose

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc - Hospital, Brussels
  - UZ Leuven, Leuven
- Tampere University Hospital, Tampere, Finland
- Germany (5):
  - Charite, Berlin
  - Universitatsklinikum Erlangen - Hospital, Erlangen
  - Universitätsklinikum Freiburg - Hospital, Freiburg im Breisgau
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz - Hospital, Mainz-GE
  - Klinikum rechts der Isa der Technischen Universitaet Muenchen - Hospital, Munich
- Netherlands (3):
  - AMC, Amsterdam
  - Ziekenhuis Rijnstate - Hospital, Arnhem
  - Maastricht University Medical Center - Hospital, Maastricht
- Norway (2):
  - Alesund Hospital, Ålesund
  - Oslo University Hospital HF, Oslo